CLINICAL TRIAL: NCT02337400
Title: Das Verhaltenstherapeutische Therapiemanual "Smoke_less" Zur Reduktion Des Tabakkonsums: Eine Evaluationsstudie Mit Ambulanten Patienten
Brief Title: Evaluation of a Cognitive Behavioral Smoking Reduction Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Oliver Pogarell, Prof. Dr. med., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eval_Smoke_less_LMU
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Tobacco Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Smoking Reduction Program (Experimental): Cognitive behavioral smoking reduction program "Smoke_less" Duration: 5 weeks with 4 weekly sessions over 2,5 hours and two phone calls
  Interventions: Behavioral: Cognitive behavioral smoking reduction program "Smoke_less"
- Counseling Interview (Active Comparator): 15 minute counseling interview
  Interventions: Behavioral: 15 minute counseling interview
- Waiting Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive behavioral smoking reduction program "Smoke_less" — Duration: 5 weeks, 4 sessions over 2,5 hours and 2 phone calls
  Arms: Smoking Reduction Program
Behavioral: 15 minute counseling interview
  Arms: Counseling Interview

SUMMARY:
The aim of this study is to evaluate a new cognitive behavioral smoking reduction program for ambulant patients in a three-armed study design. Study participants will be randomized to one of the following three study groups: experimental group: 5-week lasting cognitive behavioral reduction program ("smoke_less"); active comparator: 15 minutes counseling interview; waiting group: no intervention.

The three follow-up measures take place after the reduction program in week 6, 17 an 29. After the finalisation of the last follow-up, participants from the active comparator and waiting group get the chance to take part at the smoking reduction program at no charge.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* Result Fagerström-Test >= 3
* Consumption of at least 10 Cig./day
* carbon monoxide >= 8 ppm
* Wish, to reduce smoking but no intention to stop smoking within the next 4 weeks
* Agreement, to resign to nicotine replacement therapy, other therapies for smoking reduction, e-cigarettes or non-smoking tobacco products during study time

Exclusion Criteria:

* severe psychiatric disorder
* severe neurologic disease
* alcohol, drug or medication abuse (acute or in anamnesis)
* severe cardiovascular disease
* severe cancer disease
* severe internal disease
* Consumption of psychopharmacological medication
* acute suicidal tendency
* pregnancy or lactation
* consumption of medication therapy for smoking reduction in the last 3 month

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of smoked cigarettes/day at 6, 17 and 29 weeks | 6, 17 and 29 weeks
Change from baseline in percentage of carbon monoxide in exhalation air at 6, 17 and 29 weeks | 6, 17 and 29 weeks

SECONDARY OUTCOMES:
Change from baseline in Fagerström Test for Nicotine Dependence at 6, 17 and 29 weeks | 6, 17 and 29 weeks
Change from baseline in Questionnaire of Smoking Urges at 6, 17 and 29 weeks | 6, 17 and 29 weeks
Change from baseline in Readiness to Change Questionnaire at 6, 17 and 29 weeks | 6, 17 and 29 weeks
Change from baseline in Process of Change Questionnaire at 6, 17 and 29 weeks | 6, 17 and 29 weeks
Change from baseline in Decisional Balance Questionnaire at 6, 17 and 29 weeks | 6, 17 and 29 weeks
Change from baseline in Self-Efficacy scale for smokers 6, 17 and 29 weeks | 6, 17 and 29 weeks
Change from baseline in knowledge and skills scale about smoking reduction at 6, 17 and 29 weeks | 6, 17 and 29 weeks
Change from baseline in stress scale at 6, 17 and 29 weeks | 6, 17 and 29 weeks
Change from baseline in health satisfaction satisfaction scale at 6, 17 and 29 weeks | 6, 17 and 29 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Psychiatry, Munich, Germany

REFERENCES:
- [Derived] Ruther T, Kiss A, Eberhardt K, Linhardt A, Kroger C, Pogarell O. Evaluation of the cognitive behavioral smoking reduction program "Smoke_less": a randomized controlled trial. Eur Arch Psychiatry Clin Neurosci. 2018 Apr;268(3):269-277. doi: 10.1007/s00406-017-0818-6. Epub 2017 Jun 14. PMID 28616772